CLINICAL TRIAL: NCT03304587
Title: Effects of Bright Light on Co-occurring Cancer-related Symptoms in Breast Cancer Survivors: A Personalized Intervention
Brief Title: Effects of Bright Light on Co-occurring Cancer-related Symptoms in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Horng-Shiuann Wu, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201703147; 1R15NR016828-01A1 (NIH)
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Polysomnography; Multicenter Studies as Topic; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm 1: Bright blue-green light (Experimental): * Bright blue-green light (~515nm; 12,000 lux) for 30 minutes once a day.
  * For those who have scores of ≤41 (evening types) on Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ), light will be delivered within 30 minutes of waking for 14 consecutive mornings. For those who receive scores of ≥59 (morning types), light will be delivered between 1900-2000 hours for 14 consecutive evenings.
  * Light therapy will be self-administered using a light visor cap
  * Each participant will make (3) overnight visits to the sleep laboratory
  * On 2 randomly selected days, the participants will wear a light meter during wake time
  Interventions: Diagnostic Test: Polysomnography (PSG); Diagnostic Test: Rectal thermistor 400 Series; Other: Bright blue-green light; Diagnostic Test: Digital foot candle datalogging light meter; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer-Fatigue; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Depression; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Physical Function; Other: Pittsburgh Sleep Quality Index (PSQI); Other: Center for Epidemiological Studies - Depression; Other: Montreal Cognitive Assessment (MoCA); Other: European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC QLQ-C30); Other: Daily Log
- Arm 2: Dim red light (Active Comparator): * Dim red light (5 lux) (control group) for 30 minutes once a day.
    --For those who have scores of ≤41 (evening types) on Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ), light will be delivered within 30 minutes of waking for 14 consecutive mornings. For those who receive scores of ≥59 (morning types), light will be delivered between 1900-2000 hours for 14 consecutive evenings.
  * Light therapy will be self-administered using a light visor cap
  * Each participant will make (3) overnight visits to the sleep laboratory --On 2 randomly selected days, the participants will wear a light meter during wake time
  Interventions: Diagnostic Test: Polysomnography (PSG); Diagnostic Test: Rectal thermistor 400 Series; Other: Dim red light; Diagnostic Test: Digital foot candle datalogging light meter; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer-Fatigue; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Depression; Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Physical Function; Other: Pittsburgh Sleep Quality Index (PSQI); Other: Center for Epidemiological Studies - Depression; Other: Montreal Cognitive Assessment (MoCA); Other: European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC QLQ-C30); Other: Daily Log

INTERVENTIONS:
Diagnostic Test: Polysomnography (PSG) — Sleep patterns will be measured by in-lab PSG following a standardized protocol. 10mm silver/silver chloride electroencephalogram (EEG) and electromyography (EMG) electrodes and 11mm silver/silver chloride electroculography (EOG) electrodes will be connected to a Nihon Kohden system, 912 model (Nihon Kohden, Irvine, CA). A standard sleep montage following the 10/20 procedure for electrode placement, left and right electrooculography referenced to the opposite mastoid and mentalis electromyography will be followed. Data will be visually scored by a polysomnographer blind to study conditions following the American Academy of Sleep Medicine (AASM) Manual.
  Other Names: PSG
Diagnostic Test: Rectal thermistor 400 Series — Nocturnal core body temperature will be measured using a rectal thermistor 400 series manufactured by YSI (Yellow Springs, OH, USA) inserted up to a depth of 7 cm. and taped in place. The thermistor will be connected to a Model 4600 thermometer (YSI, Yellow Springs, OH, USA) that will be interfaced with the PSG via cabling. Core temperature readings will be continuously monitored and recorded every 5 minutes during the all-night sleep studies.
Other: Bright blue-green light — -The cap visor-mounted device controls the distance of the light exposure, and positions the light source above eye level to target on the lower retina for better effect
  Arms: Arm 1: Bright blue-green light
Other: Dim red light — -The cap visor-mounted device controls the distance of the light exposure, and positions the light source above eye level to target on the lower retina for better effect
  Arms: Arm 2: Dim red light
Diagnostic Test: Digital foot candle datalogging light meter — On 2 random days during the 2-week bright light treatment, ambient light will be recorded continuously during waking hours using a digital foot candle datalogging light meter (Extech Instruments, Waltham, MA) Model SDL400. The 7.1" x 2.9" x 1.0" light meter (12.21 oz) has the capacity to measure up to 10,000 footcandles (accuracy: ± 4% reading). The light-weight light sensor is approximately 2 inches in diameter and comes with a clip and strap that makes it comfortable to wear just below the neck.
Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer-Fatigue — 8 items with a 5-point rating scale (1=not at all to 5 =very much) measuring fatigue experience and fatigue impact. Higher scores indicate worse fatigue. PROMIS-Fatigue was developed based on rigorous methodologies. The psychometric properties have been established across chronic illnesses including cancer.
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores means more the attribute to be measures: e.g., for fatigue, sleep disturbance, depression, higher scores mean worse fatigue, worse sleep disturbance, worse depression.
  But for physical function, higher scores mean better functioning.
  Other Names: PROMIS-Cancer-Fatigue
Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep Disturbance — 8 items with 5-point rating scales measuring overall sleep and sleep-related impairments. Higher scores indicate worse sleep disturbances. Validity was supported by moderate to high correlations with the existing scales, e.g. PSQI, Epworth Sleepiness Scale (ESS). The scores significantly differed participants with and without sleep disorders.
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores means more the attribute to be measures: e.g., for fatigue, sleep disturbance, depression, higher scores mean worse fatigue, worse sleep disturbance, worse depression.
  But for physical function, higher scores mean better functioning.
  Other Names: PROMIS-Sleep Disturbance
Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Depression — 8 items with 5-point rating scales (1=never to 5=always) measuring affective and cognitive manifestations of depressive mood. Higher scores indicate worse depression. In a sample of depressed outpatients, PROMIS-Depression showed greater reliability when compared to the CES-D and the Patient Health Questionnaire (PHQ-9). Convergent validity with the CES-D and PHQ-9 was supported by strong correlations, ranged 0.72 to 0.84
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores means more the attribute to be measures: e.g., for fatigue, sleep disturbance, depression, higher scores mean worse fatigue, worse sleep disturbance, worse depression.
  But for physical function, higher scores mean better functioning.
  Other Names: PROMIS-Depression
Other: Patient-Reported Outcomes Measurement Information System (PROMIS)-Physical Function — 8 items with 5-point rating scales measuring the individual's ability to complete daily activities. Higher scores indicate worse functioning. Validity was tested in 1,415 adults with diverse clinical conditions. The PROMIS Physical Function scores corresponded to the expected positive or negative changes in the individual's physical function.
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores means more the attribute to be measures: e.g., for fatigue, sleep disturbance, depression, higher scores mean worse fatigue, worse sleep disturbance, worse depression.
  But for physical function, higher scores mean better functioning.
  Other Names: PROMIS-Physical Function
Other: Pittsburgh Sleep Quality Index (PSQI) — 19 self-report items measuring sleep quality, latency, duration, efficiency, disturbance, medication use, and daytime dysfunction. Each item is rated on a 0-3 rating scale. The global PSQI score ranges 0-21, with higher scores indicating more severe sleep disturbance. A global PSQI score greater than 5 was found to have a sensitivity of 89.6% and a specificity of 86.5% in differentiating good and poor sleepers.
  Other Names: PSQI
Other: Center for Epidemiological Studies - Depression — 20-item self-report instrument commonly used to measure depressive symptoms in cancer patients. Each item is rated on a 4-point rating scale (0=rarely or none of the time to 3=all of the time) describing the frequency of occurrence during the past week. Score can range from 0-60, with higher scores indicating more depressive symptoms.
  Other Names: CES-D
Other: Montreal Cognitive Assessment (MoCA) — The MoCA is highly sensitive for screening patient with mild cognitive impairment. The MoCA is a 30-point scale with 7 cognitive subtests: visuo-executive, naming, attention, language, abstraction, delayed recall, and orientation. It scores from 0 to 30, where higher scores indicate better cognition and a score below 26 indicates cognitive impairment. The MoCA is highly sensitive for screening patient with mild cognitive impairment.
  Other Names: MoCA
Other: European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC QLQ-C30) — The EORTC QLQ-C30 consists of 30 items with a 4-point rating scale (1=not at all to 4=very much) measuring functioning, symptom intensity, and global health status/quality of life during the past week.
  Other Names: EORTC QLQ-C30
Other: Daily Log — -A log where the participants will indicate date, wake time, sleep time answer 3 questions regarding the previous nights sleep (answers range from 1=not at all to 5=very much), have an area to indicate if naps occurred during the day, and 2 questions about fatigue & sleepiness (answers ranging from 0=no fatigue/sleepiness to 10=worst fatigue/sleepiness

SUMMARY:
This study will implement therapeutic bright light that is tailored to the individual's circadian typology and will estimate its effects on circadian rhythms, 4 common cancer-associated symptoms, and impact on quality of life in survivors living with cancer. Examining a selected phase marker (core body temperature) in relation to the associated clinical features (symptoms) is the starting point for future investigation of the biological mechanisms of symptoms.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the feasibility of implementing a home-based, personalized bright light intervention, and to estimate the effects of bright light on 4 common long-term or late effects of cancer (sleep disturbance, fatigue, depression, cognitive dysfunction) and on quality of life in post-treatment survivors of breast cancer. The three specific aims include:

Aim #1: To assess the feasibility of implementing a home-based, personalized bright light intervention and the proposed data collection plan in post-treatment survivors of breast cancer.

Aim #2: To estimate the effects of the personalized bright light intervention on sleep disturbance, fatigue, depression, cognitive dysfunction, and quality of life in survivors of breast cancer.

Aim #3: To estimate the effects of a personalized bright light intervention on circadian rhythms in survivors of breast cancer.

The participants of this randomized, controlled pilot study will be randomized to either 30-minute blue-green light therapy at 12,000 lux or dim red light control at 5 lux. Light will be self-administered using a light visor cap at home for 14 consecutive days. Tailored to the individual's circadian pattern, light will be delivered either within 30 minutes of waking in the morning or between 1900-2000 hours in the evening. The nocturnal sleep patterns will be monitored by all-night in-lab polysomnography; sleep quality, fatigue, depression, and quality of life will be self-reported; cognition will be objectively assessed before and after the intervention. Circadian rhythm will be indexed by nocturnal core body temperature before and after the intervention. Feasibility will be determined by the proportion of contacted, recruited, and retained subjects, and completeness of the data collected. Subjective feedback and burden will be assessed at study exit.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 21 years of age or older 1-3 years post-completion of chemotherapy or/and radiation therapy for stage I-III breast cancer
* Experience ≥ 2 concurrent symptoms (fatigue, sleep disruption, depressive symptoms, and/or cognitive dysfunction as measured by 4 screening instruments)
* Be either phase advanced or delayed (morning or evening types by the Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ) ≥59 or ≤41)
* Sighted
* Mentally competent to consent
* Able to understand English.

Exclusion Criteria:

* Undergoing cancer treatment for another malignancy
* Have metastatic cancer
* Engaged in shift work or travel across more than three time zones within 2 weeks prior to study
* Current diagnosis of seasonal affective disorder or substance abuse Current diagnosis of major Axis I psychiatric disorders (e.g. depressive disorders), neurological impairments, or muscular dystrophies
* Report severe depressive mood (Center for Epidemiological Studies Depression Scale (CES-D) >24)
* Take prescribed sedative hypnotics or steroids Have eye conditions (glaucoma or retinal disease), problems triggered by bright light (e.g., migraine), or take photosensitizing medications (e.g., some porphyrin drugs, antipsychotics, antiarrhythmic agents)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Shiuann Wu, PhD, Study Chair — Michigan State University College of Nursing
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu HS, Gao F, Davis JE, Given CW. Effects of chronotype-tailored bright light intervention on post-treatment symptoms and quality of life in breast cancer survivors. Support Care Cancer. 2023 Nov 17;31(12):705. doi: 10.1007/s00520-023-08157-9. PMID 37975923
- [Derived] Wu HS, Gao F, Davis JE, Given CW. Effects of Chronotype-tailored Bright Light Intervention on Symptoms and Quality of Life in Breast Cancer Survivors. Res Sq [Preprint]. 2023 Aug 25:rs.3.rs-3286350. doi: 10.21203/rs.3.rs-3286350/v1. PMID 37674711
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants withdrew prior to assignment for: schedule coordination issues (n=8); loss of contact after 3 attempts (n=2)
Groups:
- Arm 1: Bright Blue-green Light: * Bright blue-green light (~515nm; 12,000 lux) for 30 minutes once a day.
  * For those who have scores of ≤41 (evening types) on Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ), light will be delivered within 30 minutes of waking for 14 consecutive mornings. For those who receive scores of ≥59 (morning types), light will be delivered between 1900-2000 hours for 14 consecutive evenings.
  * Light therapy will be self-administered using a light visor cap
  * Each participant will make (3) overnight visits to the sleep laboratory
  * On 2 randomly selected days, the participants will wear a light meter during wake time
  Bright blue-green light: -The cap visor-mounted device controls the distance of the light exposure, and positions the light source above eye level to target on the lower retina for better effect
  **See study protocol for measurement details
- Arm 2: Dim Red Light: -Dim red light (5 lux) (control group) for 30 minutes once a day.
  * For those who have scores of ≤41 (evening types) on Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ), light will be delivered within 30 minutes of waking for 14 consecutive mornings. For those who receive scores of ≥59 (morning types), light will be delivered between 1900-2000 hours for 14 consecutive evenings.
    * Light therapy will be self-administered using a light visor cap
    * Each participant will make (3) overnight visits to the sleep laboratory
  * On 2 randomly selected days, the participants will wear a light meter during wake time
  Dim red light: -The cap visor-mounted device controls the distance of the light exposure, and positions the light source above eye level to target on the lower retina for better effect
  **See study protocol for measurement details
Period: Overall Study
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Started | 15 | 15
Withdrawal | 1 | 1
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Headache after intervention | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (8.1) | 54.2 (8.7) | 52.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Greater Lansing, Michigan | 11 | 11 | 22
  United States: St Louis Metro., Illinois/Missouri | 4 | 4 | 8
Education [Mean (Standard Deviation); unit: years] | 15.6 (2.7) | 16.5 (2.6) | 16.1 (2.7)
Marital Status [Number; unit: Participants]
  Single | 1 | 1 | 2
  Married/Partnered | 11 | 9 | 20
  Divorced | 3 | 4 | 7
  Widowed | 0 | 1 | 1
Employment [Number; unit: Participants]
  Full time | 9 | 10 | 19
  Part time | 1 | 1 | 2
  Self employed | 4 | 1 | 5
  Retired | 1 | 3 | 4
Living Arrangement [Number; unit: participants]
  Lives alone | 1 | 2 | 3
  Lives with others | 14 | 13 | 27
Tumor Stage [Number; unit: participants] — Stage I is earliest stage for most types of invasive breast cancer (ie spread to nearby tissue). Most stage I tumors are 2 centimeters or smaller.
  Stage II has not spread to distant sites, further classified depending on tumor size and any spread to lymph nodes - under arm and/or near breastbone. Even if there is no spread cancer is often classified as stage II if tumor is larger than 2 cm.
  Stage III is all inflammatory breast cancer. Also may include larger tumors and/or advanced lymph node spread. Cancer that has grown into the chest wall or breast skin is considered stage III.
  participants
    Stage I | 8 | 11 | 19
    Stage II | 5 | 3 | 8
    Stage III | 2 | 1 | 3
Previous Treatment [Number; unit: participants]
  Chemotherapy | 2 | 1 | 3
  Radiation | 8 | 10 | 18
  Both (chemotherapy & radiation) | 5 | 4 | 9
Number of Comorbidities [Number; unit: participants]
  0 | 7 | 6 | 13
  1 | 5 | 3 | 8
  2 | 3 | 3 | 6
  3 or more | 0 | 3 | 2
Chronotype [Number; unit: Participants] — Circadian chronotype (morningness, eveningness) is an individual's natural propensity for sleep/wake timing that stems from the period of endogenous circadian rhythms relative to 24-hour day/night cycle. Circadian timing differences likely contribute to variability in response to bright light therapy.
  Chronotype was based on Horne-Ostberg Morningness-Eveningness Questionnaire (MEQ). Eveningness chronotypes were those with MEQ ≤41.Morningness chronotypes were those with MEQ ≥59. Individuals with intermediate types (MEQ 42-58) were excluded from study.
  Participants
    Eveningness | 4 | 4 | 8
    Morningness | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Study Attrition and Adherence
Description: Study participants kept a daily log where they listed the dates and times they used the light visor - noting time they put it on, and the time they took it off. The light exposure were recorded to assess adherence to the treatment protocol.
  Adherence: percentage that the study participant used the light visor for 30 minutes per day during the 14-day light therapy intervention (based on the daily log that reported use or not use of the light visor for 30 minutes for the 14 days of the intervention and the time they put it on each day and took it off each day)
  Attrition: study participants withdrew from the study prior to completing the intervention
Time Frame: Up to 3 weeks from registration
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
Participants
  Attrition | 1 | 1
  Adherence to light therapy | 14 | 14

2. Secondary Outcome: Effects of Bright Light on Sleep Disturbance as Measured by the PROMIS-Sleep Disturbance
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-Sleep disturbance T-Score.
  A higher PROMIS-Sleep disturbance T-score represents greater\worse sleep disturbance.
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores mean worse sleep disturbance
  Note: For negatively-worded concepts like Fatigue, a T-score of 60 is one SD worse than average. By comparison, a Fatigue T-score of 40 is one SD better than average.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
T-score
  Baseline | 56 (6) | 57.3 (7.5)
  Post-Test | 49.6 (5.3) | 50.4 (6)

3. Secondary Outcome: Effects of Bright Light on Sleep Disturbance as Measured by the PSQI
Description: Pittsburgh Sleep Quality Index (PSQI) Global score:
  The PSQI has 7 components, with each component self-rated from 0-3, with 3 being worse sleep quality. Global PSQI sleep score is the sum of all 7 components, with score range from 0-21, with higher score meaning worse sleep quality.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 9.3 (3.2) | 9.6 (3.2)
  Post-Test | 7.8 (2.4) | 6.0 (3.1)

4. Secondary Outcome: Effects of Bright Light on Fatigue as Measured by the PROMIS-Cancer-Fatigue
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer-Fatigue T-Score.
  A higher PROMIS-Cancer-Fatigue T-score represents greater\worse fatigue.
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores mean worse fatigue
  Note: For negatively-worded concepts like Fatigue, a T-score of 60 is one SD worse than average. By comparison, a Fatigue T-score of 40 is one SD better than average.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
T-score
  Baseline | 55.8 (6.8) | 56.3 (7.9)
  Post Test | 48.3 (4.4) | 50.5 (6.4)

5. Secondary Outcome: Effects of Bright Light on Fatigue as Measured by the Daily Log
Description: Fatigue self-report is rated numerically from 1-5, with greater score meaning more fatigue
Time Frame: Kept throughout the approx 3 weeks of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline self-reported fatigue | 3.54 (2.03) | 4.57 (2.41)
  Post-Test self-reported fatigue | 1.92 (1.44) | 2.86 (2.35)

6. Secondary Outcome: Effects of Bright Light on Depression as Measured by the PROMIS-Depression
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-Depression T-Score.
  A higher PROMIS-Depression T-score represents greater\worse Depression.
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores mean worse worse depression.
  Note: For negatively-worded concepts like Fatigue, a T-score of 60 is one SD worse than average. By comparison, a Fatigue T-score of 40 is one SD better than average.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
T-score
  Baseline | 50.4 (7.9) | 51.1 (6.4)
  Post-Test | 45.2 (5.9) | 46.5 (7.0)

7. Secondary Outcome: Effects of Bright Light on Depression as Measured by the CES-D
Description: Center for Epidemiologic Studies Depression Scale (CES-D) score:
  Total CES-D range is 0-60, with higher score meaning more depressed.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 14.7 (8.3) | 16.3 (4.1)
  Post-Test | 6.0 (3.8) | 8.9 (5.3)

8. Secondary Outcome: Effects of Bright Lights on Cognitive Dysfunction as Measured by the MoCA
Description: MoCA (Montreal Cognitive Assessment):
  Test conducted by researcher, with total score range 0-30. Higher score means less cognitive dysfunction.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline | 27.9 (1.7) | 26.6 (2.2)
  Post-Test | 28.0 (2.0) | 27.1 (1.7)

9. Secondary Outcome: Effect of Bright Light on Quality of Life as Measured by the PROMIS-Physical Function
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-Physical Function T-Score.
  A higher PROMIS-Physical Function T-score represents greater\better Physical Function.
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). A mean of 50 equals the mean in the U.S. general population.
  Higher scores mean better functioning.
  Note: A T-score of 60 is one SD greater than average; A T-Score of 40 is one SD lower than average.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
T-score
  Baseline | 47.5 (10.2) | 48.6 (8.1)
  Post-Test | 48.7 (9.2) | 51.3 (8.3)

10. Secondary Outcome: Effect of Bright Light on Quality of Life as Measured by EORTC QLQ-30
Description: Quality of Life (QOL)-Global Health score: Range 0-100, higher score is better global health quality of life Quality of Life (QOL) Symptom score: Range 0-100, Higher score is worse symptoms quality of life Quality of Life (QOL)-Function: Range 0-100, Higher score is better functional quality of life
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
score on a scale
  Baseline QOL-Global | 65.6 (16.6) | 76.1 (16.0)
  Post-Test QOL-Global | 76.2 (7.9) | 81.0 (11)
  Baseline QOL-Symptom | 20.7 (13.0) | 19.5 (9.0)
  Post-Test QOL-Symptom | 13.4 (7.1) | 12.1 (7.3)
  Baseline QOL-Function | 76.7 (15.7) | 80.4 (10.4)
  Post-Test QOL-Function | 87.0 (6.6) | 87.6 (9.2)

11. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-Total Sleep Time
Description: Objective testing using in-lab polysomnography (PSG) is used to measure the effects of bright light on level of stress. Minutes of total sleep time is reported.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
minutes
  Baseline | 394.2 (68.9) | 393.53 (59.35)
  Post-Test | 386.1 (84.8) | 415.9 (71.5)

12. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-Sleep Efficiency
Description: Objective testing using in-lab polysomnography (PSG)is used to measure the effects of bright light on level of stress. Sleep efficiency is reported as percentage of total sleep time.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
percentage of sleep time
  Baseline | 81.9 (7.9) | 82.7 (8.08)
  Post-Test | 81.0 (14.3) | 82.4 (12.2)

13. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-Sleep Onset Latency
Description: Objective testing using in-lab polysomnography (PSG) is used to measure the effects of bright light on level of stress. Minutes of latency to sleep onset is reported.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
minutes
  Baseline | 58.6 (64.8) | 43.9 (49.5)
  Post-Test | 35.7 (33.1) | 52.4 (55.4)

14. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-Awakenings
Description: Objective testing using in-lab polysomnography (PSG)is used to measure the effects of bright light on level of stress. Minutes of awakenings during sleep is recorded.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
minutes
  Baseline | 20.5 (8.6) | 16.4 (7.1)
  Post-Test | 15.6 (5.2) | 15.2 (6.0)

15. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-Arousals
Description: Objective testing using in-lab polysomnography (PSG)is used to measure the effects of bright light on level of stress. Arousal minutes during sleep are recorded
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
minutes
  Baseline | 53.4 (20.4) | 64.6 (40.7)
  Post-Test | 45.8 (17.9) | 58.0 (32.2)

16. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-Arousal Index
Description: Objective testing using in-lab polysomnography (PSG) is used to measure the effects of bright light on level of stress. Arousal index is total number of arousals per hour of sleep.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: Total number of arousals per hr of sleep
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
Total number of arousals per hr of sleep
  Baseline | 8.4 (3.5) | 9.6 (5.3)
  Post-Test | 7.8 (2.8) | 8.1 (4.0)

17. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-Wake After Sleep Onset (WASO)
Description: Objective testing using in-lab polysomnography (PSG) is used to measure the effects of bright light on level of stress. Minutes till wake after sleep onset is reported.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
minutes
  Baseline | 51.6 (19.9) | 47.8 (22.7)
  Post-Test | 72.8 (41.5) | 48.2 (31.4)

18. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-sleep Stages (Min)
Description: Objective testing using in-lab polysomnography (PSG) used to measure effects of bright light on level of stress. Minutes spent in each sleep stage is reported.
  Stage 1 is when a person first falls asleep, normally lasts 1-7minutes. Body has not fully relaxed, though body and brain activities start to slow with periods of brief movements.
  Stage 2 the body enters a more subdued state including a drop in temperature, relaxed muscles and slowed breathing and heart rate.
  Stage 3 muscle tone, pulse and breathing rate decrease as body relaxes. REM brain activity picks up, body experiences atonia-a temporary paralysis of muscles except for eyes and muscles that control breathing. Usually takes 90 minutes to reach REM stage.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
minutes
  Baseline Stage 1 | 26.0 (12.6) | 28.2 (13.9)
  Post-Test Stage 1 | 24.7 (7.9) | 26.1 (14.5)
  Baseline Stage 2 | 236.7 (49.1) | 241.2 (55.4)
  Post-Test Stage 2 | 250.3 (61.3) | 279.9 (74.3)
  Baseline Stage 3 | 37.7 (40.0) | 32.5 (23.4)
  Post-Test Stage 3 | 27.1 (30.2) | 23.4 (27.4)
  Baseline REM | 93.9 (30.7) | 91.7 (28.9)
  Post-Test REM | 84.0 (28.9) | 86.5 (33.9)

19. Secondary Outcome: Effects of Bright Light on Level of Stress as Measured by the PSG-sleep Stages (%)
Description: Objective testing using in-lab polysomnography (PSG) is used to measure the effects of bright light on level of stress. Percentage of time in each sleep stage is reported.
  Stage 1 is when a person first falls asleep, normally lasts 1-7minutes. Body has not fully relaxed, though body and brain activities start to slow with periods of brief movements.
  Stage 2 the body enters a more subdued state including a drop in temperature, relaxed muscles and slowed breathing and heart rate.
  Stage 3 muscle tone, pulse and breathing rate decrease as body relaxes. REM brain activity picks up, body experiences atonia-a temporary paralysis of muscles except for eyes and muscles that control breathing. Usually takes 90 minutes to reach REM stage.
Time Frame: Baseline (day 2 of study) and Post-treatment (approx day 17 of study)
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
Number analyzed (Participants) | 15 | 15
percentage of sleep time
  Baseline Stage 1 | 6.9 (4.0) | 7.4 (4.4)
  Post-Test Stage 1 | 6.7 (2.9) | 6.3 (3.3)
  Baseline Stage 2 | 60.6 (10.7) | 61.0 (7.7)
  Post-Test Stage 2 | 64.8 (7.7) | 66.7 (11.0)
  Baseline Stage 3 | 9.2 (9.0) | 8.5 (6.6)
  Post-Test Stage 3 | 7.3 (7.5) | 6.4 (8.4)
  Baseline REM | 23.4 (5.4) | 23.2 (6.5)
  Post-Test REM | 21.2 (5.8) | 20.7 (6.9)

ADVERSE EVENTS:
Time Frame: Baseline assessment through post-assessment (up to 3 weeks)
Description: Self-reported symptoms following intervention
Arm/Group | Arm 1: Bright Blue-green Light | Arm 2: Dim Red Light
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Bright Blue-green Light (N=15) | Arm 2: Dim Red Light (N=15)
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Participant self-report of headache following intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03304587/Prot_003.pdf
  • Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03304587/SAP_004.pdf
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT03304587/ICF_005.pdf